

## NON-INTERVENTIONAL (NI) STUDY PROTOCOL

#### **Study information**

| Title | Comparing Patient-Reported Outcomes Between Rimegepant and Triptan Users with Migraine in the United States |
|---|---|
| Protocol number | C4951076 |
| Protocol version identifier | 1.0 |
| Date | 04 October 2024 |
| Active substance | Analgesics, calcitonin gene-related peptide (CGRP) antagonists. ATC code: N02CD06 |
| Medicinal product | Rimegepant (Nurtec 75mg ODT) |
| Research question and objectives | The goal of this research is to assess patient-reported outcomes (PROs), specifically treatment satisfaction, healthcare resource use (HCRU), quality of life (QoL), work productivity loss, and migraine-specific disability of Rimegepant users, relative to triptan users, among US adults diagnosed with migraine. Secondarily, a sensitivity analysis will be conducted, applying a more restrictive definition for the Rimegepant acute user cohort, to corroborate the initial set of results. Findings from these analyses may be used to inform communications with payers regarding reimbursement of Rimegepant. |
| <b>Country of study</b> | United States (US) |
| Author | PPD |

This document contains confidential information belonging to Pfizer. Except as otherwise agreed to in writing, by accepting or reviewing this document, you agree to hold this information in confidence and not copy or disclose it to others (except where required by applicable law) or use it for unauthorized purposes. In the event of any actual or suspected breach of this obligation, Pfizer must be promptly notified.

#### 1. TABLE OF CONTENTS

| 1. TABLE OF CONTENTS | 2 |
|---|---|
| 2. LIST OF ABBREVIATIONS | 4 |
| 3. RESPONSIBLE PARTIES | 6 |
| 4. ABSTRACT | 7 |
| 5. AMENDMENTS AND UPDATES | 8 |
| 6. MILESTONES | 9 |
| 7. RATIONALE AND BACKGROUND | 9 |
| 8. RESEARCH QUESTION AND OBJECTIVES | 10 |
| 9. RESEARCH METHODS | 10 |
| 9.1. Study Design | 10 |
| 9.2. Setting | 10 |
| 9.2.1. Inclusion Criteria | 10 |
| 9.2.2. Exclusion Criteria | 11 |
| 9.3. Variables | 11 |
| 9.4. Data Sources | 14 |
| 9.5. Study Size | 14 |
| 9.6. Data Management | 15 |
| 9.7. Data Analysis | 15 |
| 9.8. Quality Control | 16 |
| 9.9. Limitations of the Research Methods | 17 |
| 9.10. Other Aspects | 17 |
| 10. PROTECTION OF HUMAN PARTICIPANTS | 17 |
| 10.1. Patient Information | 17 |
| 10.2. Patient Consent | 17 |
| 10.3. Institutional Review Board (IRB)/ Independent Ethics Committee (IEC) | 17 |
| 10.4. Ethical Conduct of the Study | 17 |
| 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS | 18 |
| 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS | |
| 13. REFERENCES | 18 |

| 14. LIST OF TABLES | 20 |
|---------------------------------------|----|
| 15. LIST OF FIGURES | 20 |
| ANNEX 1. LIST OF STANDALONE DOCUMENTS | 20 |
| ANNEY 2 ADDITIONAL INFORMATION | 20 |

#### 2. LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|--------------|--------------------------------------------|
| AAN | American Academy of Neurology |
| AE | Adverse event |
| ATT | Average treatment effect of treated |
| CGRP | Calcitonin gene-related peptide |
| ER | Emergency room |
| FDA | Food and Drug Administration |
| GCS | Global composite score |
| HCRU | Health care resource use |
| HRQoL | Health related quality of life |
| IEC | Independent ethics committee |
| IP | Internet Protocol |
| IPTW | Inverse probability of treatment weighting |
| IRB | Institutional review board |
| mAb | Monoclonal Antibody |
| MCS | Mental composite score |
| MIDAS | Migraine Disability Assessment Scale |
| NHWS | National Health and Wellness Survey |
| NSAID | Non-steroidal anti-inflammatory drugs |
| OLS | Oracle Life Sciences |
| OTC | Over the counter |
| PCS | Physical composite score |
| PRO | Patient-reported outcome |
| QoL | Quality of life |

| US | United States of America |
|---------|------------------------------------------------------------|
| WPAI-GH | Work Productivity and Activity Impairment – General Health |

#### 3. RESPONSIBLE PARTIES

### Principal Investigator(s) of the Protocol

| Name, Degree(s) | Job Title | Affiliation | Address |
|---|---|---|---|
| Simon Dagenais, PhD | Evidence Generation | Pfizer Inc | 1 Portland St, Cambridge, MA |
| | Innovation Lead | | 02139 |
| Martine C. Maculaitis, | Sr. Evidence Generation | Oracle Life Sciences | 2300 Oracle Way Austin, TX |
| PhD, MA | Lead, Real World | | 78741 USA |
| | Evidence | | |

## Additional Investigator(s) of the Protocol

| Name, Degree(s) | Job Title | Affiliation | Address |
|---|---|---|---|
| PPD | PPD | Pfizer Inc | 66 Hudson Blvd E, Fl 20, New<br>York, NY 10001 USA |
| PPD | | Pfizer Inc | 1 Portland St, Cambridge, MA<br>02139 |
| PPD , MPH, PhD | | Oracle Life Sciences | 2300 Oracle Way Austin, TX<br>78741 USA |
| PPD | | Oracle Life Sciences | 2300 Oracle Way Austin, TX<br>78741 USA |

## 4. ABSTRACT

None.

#### 5. AMENDMENTS AND UPDATES

None.

#### 6. MILESTONES

Minimum requirements:

| Milestone | Planned Date |
|-------------------------------|------------------|
| Initiation of data analysis | 05 October 2024 |
| First draft of abstract | 10 October 2024 |
| Final abstract | 15 October 2024 |
| Completion of data analysis | 20 November 2024 |
| First draft of poster content | 01 March 2025 |
| Final poster content | 15 March 2025 |

#### 7. RATIONALE AND BACKGROUND

Triptans, also known as serotonin receptor agonists, are considered as a standard treatment for acute migraine and have been widely prescribed in the United States <sup>1</sup>. A systematic review showed that standard dose (taken orally or intranasally) of triptans alleviated pain within 2 hours in 42 to 76% of patients and provided sustainable headache relief at 24 hours in 29% to 50% of patients <sup>2</sup>. However, triptans are not for preventing migraine and are associated with numerous adverse events including nausea, dizziness, and coronary vasoconstriction <sup>3</sup>.

Rimegepant, an oral medication which works by blocking the calcitonin gene-related peptide (CGRP) receptors, was approved by the Food and Drugs Administration (FDA) in February 2020, as an alternative method for the acute treatment of migraine in adults <sup>4</sup>. Rimegepant relieves pain as well as incommodious symptoms and can prevent migraine when given the proper dose <sup>5</sup>. However, nausea, urinary tract infection, and dizziness were adverse events reported for Rimegepant <sup>6</sup>.

Both triptans and Rimegepant are commonly prescribed for acute migraine but have different efficacy and side effects. Triptans showed better pain relief compared to gepants, whereas gepants were associated with fewer adverse events compared with triptans  $^1$ . Recent research also showed Rimegepant being more effective in the acute treatment of migraine in adults with a history of insufficient response to 1 or  $\ge 2$  triptans among and in current triptan users  $^7$ .

As patients with migraine tend to experience worse health status, reduced health-related, reduced work productivity, the impact of treatment in improving patient reported outcomes is critical <sup>8,9</sup>. Among triptan users, the HRQoL and work productivity were significantly impacted in those with insufficient response to triptans <sup>10</sup>. In addition to the reduction in migraine frequency, Rimegapant was associated with improvement in HRQoL over time <sup>11</sup>. However, few studies have comprehensively examined patient reported outcomes among Rimegepant users compared with triptan users. As such, the purpose of this study was to assess patient-reported outcomes (PROs) including treatment satisfaction, healthcare

resource use (HCRU), quality of life (QoL), work productivity loss, and migraine-specific disability of Rimegepant users, relative to triptan users.

#### 8. RESEARCH QUESTION AND OBJECTIVES

The primary aim of this analysis is to assess PROs, specifically treatment satisfaction, HCRU, QoL, work productivity loss, and migraine-specific disability of Rimegepant users, relative to triptan users, among US adults diagnosed with migraine.

Secondarily, a sensitivity analysis will be conducted, applying a more restrictive definition for the Rimegepant user cohort, to corroborate the initial set of results. Findings from these analyses may be used to inform communications with payers regarding reimbursement of Rimegepant.

#### 9. RESEARCH METHODS

#### 9.1. Study Design

This is a cross-sectional study using the 2023 US (N=75,007) National Health and Wellness Survey (NHWS) data. People who use Rimegepant will be compared with those who use triptan on treatment satisfaction, HCRU, QoL, work productivity loss, and migraine-specific disability outcomes. The cross-sectional design allows us to compare the Rimegepant vs. triptan users on multiple outcomes in a relatively quick and inexpensive way.

#### 9.2. Setting

All data from the NHWS are reported by the respondent. NHWS participants are recruited through an existing, general-purpose (i.e., not health care-specific) web-based consumer panel via opt-in e-mails, co-registration with panel partners, e-newsletter campaigns, banner placements, and affiliate networks. All panelists explicitly agree to be a panel member, register with the panel through a unique e-mail address, and complete an in-depth demographic registration profile. A stratified random sampling procedure is implemented to ensure that the demographic composition of the final NHWS sample is representative of the general adult population in the US. In each year the NHWS is fielded, data from the International Database of the US Census Bureau are used to identify the relative proportions of adults by age, race/ethnicity, and gender; these proportions are then mimicked during the recruiting of panel members.

#### 9.2.1. Inclusion Criteria

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

- 1. Patients who have consented to the anonymous use of their data for research purpose.
- 2. Aged 18 or older.
- 3. Self-reported a diagnosis of migraine by physician.
- 4. Currently on Rimegepant or triptan (via oral route) use at time of survey.

- 5. In addition, patients to be included in the sensitivity analysis need to meet the following criteria:
  - Currently on acute Rimegepant use (<12 days using Rimegepant per month), or triptan (via oral route) use at time of survey.

#### 9.2.2. Exclusion Criteria

Patients meeting the following criteria will not be included in the study:

1. Currently on both Rimegepant and triptan use at time of survey.

#### 9.3. Variables

The NHWS includes self-reported data on demographics, health characteristics, disease history, and health outcomes. The Table 1 below provides further details on the specific variables that will be assessed in the study.

**Table 1. Study Variables** 

| Variable | Role | Operational Definition |
|---|---|---|
| Rimegepant vs. triptan | Exposure | Current Rimegepant users (for sensitivity analysis |
| use | | restricted to acute Rimegepant users with <12 days use per |
| | | month) vs. triptan users (no OTC, oral route only). |
| Outcomes: Migraine trea | Outcomes: Migraine treatment use and treatment satisfaction | |
| Migraine medication | Outcome | Defined as drug only, OTC only and both drug and OTC, |
| type (drug or OTC) | | based on current use of migraine medication classes |
| Migraine treatment type | Outcome | Defined as acute only, prevention only and both acute and |
| (acute or prevention) | | prevention, based on current use of migraine medication classes |
| Total number of acute | Outcome | Total number of acute agent classes (both drug and OTC) |
| migraine agent drug | | used |
| (continuous) | | |
| Total number of acute | Outcome | Including 1 drug class, 2 or more drug classes, and 3 or |
| migraine agent drug | | more drug classes based on the total number of acute |
| (categorical) | | agent (both drug and OTC) classes used |
| Total number of | Outcome | Total number of prevention agent classes (only drug) used |
| prevention migraine | | |
| agent drug (continuous) | | |
| Total number of | Outcome | Including 1 drug class, 2 or more drug classes, and 3 or |
| prevention migraine | | more drug classes based on the total number prevention |
| agent drug (categorical) | | agent classes (only drug) used |
| Current migraine | Outcome | Defined as yes or no for current migraine treatments on |
| treatments (drugs) | | drug classes including: Rimegepant, triptans, NSAIDs, |
| | | opioids, barbiturates, ergots, gepants (acute, including |
| | | Rimegepant), ditan, combination analgesics, other acute |
| | | drugs, anticonvulsants, beta-blocker, antidepressant, |
| | | CGRP mAb, botox, and gepant (prevention, including Rimegepant) |
| Treatment satisfaction | Outcome | Treatment satisfaction of drug classes of: Rimegepant, all |
| (drugs) | Outcome | acute agents, triptans, NSAIDs, opioids, barbiturates, |
| (urugo) | | ergots, gepants (acute), ditans, combination analgesics, |
| | | other acute treatment, all prevention agents, |
| | | other acute treatment, an prevention agents, |

| | | 1 |
|---|---|---|
| | | anticonvulsants, beta-blockers, antidepressants, CGRPs mAb, botox, and gepant (prevention) Categorized into 7 categories: extremely dissatisfied, very dissatisfied, somewhat dissatisfied, neither dissatisfied nor satisfied, somewhat satisfied, very satisfied, extremely satisfied |
| Current migraine treatments (OTC) | Outcome | Defined as yes or no for current migraine treatments on OTC classes of analgesics (acetaminophen only), analgesics (combinations), NSAIDs, other OTCs |
| Treatment satisfaction-<br>analgesics<br>(acetaminophen only) | Outcome | Treatment satisfaction of OTC classes of analgesics (acetaminophen only), analgesics (combinations), NSAIDs, and other OTCs Categorized into 7 categories: extremely dissatisfied, very dissatisfied, somewhat dissatisfied, neither dissatisfied nor satisfied, somewhat satisfied, very satisfied, extremely satisfied |
| Outcomes: HRQoL | | |
| RAND-36<br>EQ-5D-5L | Outcome Outcome | PCS, MCS, and GCS index scores of the RAND-36 <sup>12</sup> Health state utilities and the EuroQoL Visual Analog |
| WPAI-GH | Outcome | Scale (EQ-VAS) <sup>13</sup> Absenteeism (% of work time missed because of one's health in the past 7 days), presenteeism (% impairment experienced while at work in the past 7 days because of one's health), overall work impairment (combination of absenteeism and presenteeism), and activity impairment (% impairment in daily activities because of one's health in the past 7 days) among total population, employed, unemployed, and disabled <sup>14</sup> |
| MIDAS | Outcome | Total score, categorical (grade I-IV), and item scores (1-7) of MIDAS <sup>15</sup> |
| Outcomes: HCRU | | |
| ER visits | Outcome | Visited ER in past 6 months (yes or no); number of ER visits in past 6 months among total population and participants with ER visits |
| Hospitalizations | Outcome | Was hospitalized in past 6 months (yes or no); number of hospitalizations in past 6 months among total population and participants with hospitalizations |
| General<br>practitioner/family<br>practitioner visits | Outcome | Visited general practitioner/family practitioner in past 6 months (yes or no); number of general practitioner/family practitioner visits in past 6 months among total population and participants with general practitioner/family practitioner visits |
| Cardiologist visits | Outcome | Visited cardiologist in past 6 months (yes or no); number of cardiologist visits in past 6 months among total population and participants with cardiologist visits |
| Neurologist visits | Outcome | Visited neurologist in past 6 months (yes or no); number of neurologist visits in past 6 months among total population and participants with neurologist visits |
| Traditional healthcare provider visits | Outcome | Visited traditional healthcare provider in past 6 months (yes or no); number of traditional healthcare provider visits in past 6 months among total population and participants with traditional healthcare provider visits |
| Covariates adjusted thr | | |
| Age (continuous) | Potential confounder | Age of participants in years |

| C | D-44:-14 | M-1 f1- |
|---|---|---|
| Sex | Potential confounder | Male vs. female |
| Race | Potential confounder Potential confounder | Categorized as black, white, and other Yes vs. no |
| Hispanic/Latino<br>Marital status | Potential confounder Potential confounder | Single/ not living with partner vs. married/ living with partner |
| Health insurance | Potential confounder | Categorized as private insurance, public insurance, no insurance, and unsure |
| University education | Potential confounder | Less than university education vs. university education or higher |
| Annual household income | Potential confounder | Categorized as below median income (<50,000), median income (\$50,000-\$74,999), above median income (≥\$75,000), and decline to answer |
| Employed | Potential confounder | Yes (full-time/ part-time/ self-employed) vs. no |
| Charlson comorbidity index | Potential confounder | Charlson comorbidity index scores with and without patients of score 0 and categories based on scores: 0, 1, 2, 3, and 4+ |
| Body mass index | Potential confounder | Body mass index in kg/m <sup>2</sup> |
| Alcohol use | Potential confounder | Currently drink alcohol vs. currently do not drink alcohol |
| Smoking status | Potential confounder | Categorized as current smoker, former smoker, and never smoked |
| Exercise | Potential confounder | Number of days exercise per months |
| Contraindications | Potential confounder | Ever experienced each of contraindications (angina, arrythmia, atrial fibrillation, congestive heart failure, heart attack, left ventricular hypertrophy, mini-stroke/transient ischemia attack, peripheral arterial disease /poor circulation, Peripheral vascular disease, stroke, and unstable angina/chest pains) |
| Cardiovascular risk factors | Potential confounder | Ever experienced each of cardiovascular risks (high blood pressure, high cholesterol, current smoker, type 2 Diabetes, and obesity) |
| Any contraindications | Potential confounder | Ever experienced any contraindications listed above |
| Any cardiovascular risk factors | Potential confounder | Ever experienced any cardiovascular risks factors listed above |
| Any contraindications or cardiovascular risk factors | Potential confounder | Ever experienced any contraindications or cardiovascular risks factors listed above |
| Time since migraine diagnosis | Potential confounder | Time since migraine diagnosis in years |
| Monthly migraine days (continuous) | Potential confounder | Number of days experienced migraine in past 30 days |
| Monthly headache days (continuous) | Potential confounder | Number of days experienced headache in the past 30 days |
| Medication overuse (migraine only) | Potential confounder | Yes or no, for migraine-specific medications only |
| | l be evaluated for balar | ice between exposure groups |
| Age (categorical)* | Potential confounder | Categorized based on age of participants in years: 18-29, 30-39, 40-49, 50-59, 60-69, 70-79, 80-89 |
| Monthly migraine days (categorical)* | Potential confounder | Categorized based on number of days experienced migraine in past 30 days: <4, 4-9, 10-14, and ≥15 |
| Monthly headache days (categorical)* | Potential confounder | Categorized based on number of days experienced headache in past 30 days: <4, 4-9, 10-14, and ≥15 |
| Experience migraines related to menstrual cycle | Potential confounder | Yes vs. no, female participants only |

\*Categorical age, monthly migraine days, and monthly headache days will be included in inverse probability of treatment weighting (IPTW) adjustment if their distributions are not balanced (standardized mean difference >0.1) after IPTW.

Abbreviations: OTC: over the counter; NSAID: non-steroidal anti-inflammatory drugs; CGRPs mAb: calcitonin gene-related peptide antibodies monoclonal antibodies; HRQoL: health related quality of life; PCS: physical composite score; MCS: mental composite score; GCS: global composite score; WPAI-GH: the Work Productivity and Activity Impairment – General Health; MIDAS: Migraine Disability Assessment Scale; HCRU: health care resource utilization; ER: emergency room; IPTW: inverse probability of treatment weighting

#### 9.4. Data Sources

This study will use self-reported data sourced from the NHWS. The NHWS is an annual, cross-sectional, internet-based survey of adults conducted across several countries annually. The current study will use data from the 2023 US (N=75,007) NHWS.

#### 9.5. Study Size

Sample size estimates, based upon preliminary feasibility, are provided below, in Table 2. The sample size for this study is fixed by the number of patients in the NHWS database who meet the imposed criteria.

**Table 2.** Estimated Sample Sizes

| Patient Cohorts | n |
|----------------------------------------------------------------|--------|
| Overall NHWS sample | 75,007 |
| Diagnosed with migraine | 8,439 |
| Triptan users (oral route only, no OTC) without Rimegepant use | |
| Rimegepant users without triptan use | |
| Rimegepant users (acute only) without triptan use* | 112 |

<sup>\*</sup>For sensitivity analysis.

Abbreviations: NHWS: National Health and Wellness Survey; OTC: over the counter

A sample size of 1) 130 and 2) 100 in each group (1:1 allocation) will have 80% power to detect an effect size of at least 1) 0.35 standard deviation (SD) units (indicative of at least a "small-to-medium" effect) and 2) 0.4 SD units (indicative of a medium effect), respectively, using a 2-group t-test with a 5% 2-sided significance level. We will have a sample size much greater than 130 in one of our groups, resulting in higher statistical power compared to the 1:1 allocation mentioned above. A total sample size of 100 will have 80% power to detect an effect size from a chi-square distribution of at least 0.33 (indicative of at least a "small-to-medium" effect) using a chi-square test with a 5% 2-sided significance level and 3 degrees of freedom. There will be sufficient power to detect a "small-to-medium" effect of Rimegepant user vs. triptan use on the outcomes in the main analysis, and sufficient power to detect a medium effect in the sensitivity analysis with acute Rimegepant users only.

#### 9.6. Data Management

This study will use previously collected data that have been deidentified, processed, and cleaned. Prior to initiating the study programming, procedures were implemented to assess the quality of responses including, but not limited to, response ranges, consistency, and skip patterns. Data entry was completed instantaneously as the respondent answered the survey questions. Therefore, there are no paper surveys to house or destroy, and no manual data entry is required. The database that houses the questionnaire responses allows for direct exportation into statistical software. Identifying information about panel members will not be released other than a single panel identification number. Therefore, the working data files contain no identifying information, apart from the panel identification number. Specifically, the dataset does not include names, addresses, or any other information that can personally identify the respondents.

Quality checks were implemented on the dataset before it became final. These checks included Internet Protocol (IP) address checks (i.e., ensuring the respondent resided within the country stated and that a single IP address was not associated with multiple panel accounts), completion times (ensuring a respondent did not complete the survey in a timeframe that was too short, implying inattentiveness), illogical/inconsistent data responses, etc. At the discretion of the data management team, respondents who failed these checks were excluded from the final dataset.

The statistical software package that will be used for the study is R 4.3.1 (R Project for Statistical Computing).

#### 9.7. Data Analysis

The average treatment effect of treated (ATT) will be measured to evaluate the effects of Rimegepant vs. triptan among current Rimegepant users.

Based on clinical relevance, we will prespecify a list of variables to adjust for the comparison.

Inverse probability of treatment weighting (IPTW) will be conducted to adjust for confounding by the covariates. The propensity score for each participant will be estimated by logistic regression and by including the prespecified list of variables to adjust for. Weights for ATT will be calculated for both exposed (Rimegepant users) and unexposed group (triptan users) <sup>16</sup>. Stabilized weights will be used to address extreme weight values.

To confirm that the IPTW procedure is successful, the weighted Rimegepant users and triptan users will be compared on the covariates using standardized mean difference (SMD) to ensure both groups are adequately balanced across all weighting criteria. While there is no definitive cut-off for identifying imbalance in IPTW, as a rule of thumb, a standardized mean difference (SMD) that is >0.10 is indicative of imbalance <sup>17</sup>. This threshold will be applied to determine the quality of the weighting.

Once the weighting is confirmed to be successful, bivariate analyses will be conducted to compare the weighted cohorts on treatment satisfaction, HCRU, QoL, migraine-specific

disability, and work productivity loss. Specifically, categorical variables will be analyzed using chi-square tests or Fisher's exact tests for small samples; continuous variables will be analyzed using 2-sample t-tests. Non-parametric tests may be considered for comparisons on skewed variables (e.g., HCRU) when the sample size is small (e.g., <30). For bivariate comparisons, p-values <0.05, 2-tailed, will be considered statistically significant. If there are covariates that are unbalanced after weighting (i.e., SMD >0.1), those covariates will be adjusted for in the regression analysis of outcomes. Generalized linear models will be fit depending on the distributions of outcomes.

As a sensitivity analysis, the aforementioned IPTW and bivariate comparisons will be replicated after restricting the Rimegepant user cohort to the subset of those presumed to be acute treatment users (<12 days using Rimegepant).

A sensitivity analysis will be conducted by incorporating NHWS sampling weights into the IPTW process. Sampling weights will be applied in the logistic regression to predict the propensity score, and the final weight will be the product of the propensity score weight and the sampling weight. Bivariate comparisons will then be replicated after using these newly derived weights for the participants.

#### 9.8. Quality Control

This is a non-interventional retrospective study, so issues of quality control at study sites, e.g., data queries, do not apply. The following programming specifications will be used:

- NHWS survey includes single select questions, multi select multiple choice questions, as well as open-ended questions (e.g., asking participants to type in the types of over-the-counter medications they were taking).
- NHWS data to be used in this study will be downloaded from the Oracle server and saved as a separate data file. This data file will be stored in a secure folder on the Oracle server, which is backed up in multiple iterations on a regular basis.
- Programming code will be created for data management. This programming code will include the creation of cohort variables or any other derived variables.
- All analyses will be performed using R 4.3.1 (R Project for Statistical Computing). For quality assurance purposes, a second independent researcher will review the programming code to be used for analysis.
- Programming code used for data management and programming code used for analysis will be stored on the Oracle server and will be backed up on a regular basis.
- Data will be reviewed for quality control prior to data analysis by OLS. For example, if a respondent entered the same number for most responses, or followed a pattern in their responses, they would be considered for removal from analysis. In addition, prior to data analysis, all variables are cleaned and checked for outliers and inconsistencies by OLS.

#### 9.9. Limitations of the Research Methods

The data from the NHWS are self-reported; thus, independent, or clinical verification of responses will not be possible. Due to the self-reported nature of the data, recall error or other response biases may potentially introduce measurement error. However, many of the measures included in the study were developed solely for the purposes of patient self-report (RAND-36, EQ-5D-5L, WPAI-GH, MIDAS), and self-report is a valid and appropriate methodology for assessing subjective outcomes. Because of the cross-sectional nature of the data, causal inferences cannot be drawn, and longitudinal fluctuations in the relationships between study variables cannot be determined. While IPTW will be used to control for potential confounders, it is possible there are other variables that could not be included in the analyses that may at least partially explain any relationships observed in the current study. Finally, while the NHWS is designed to reflect the demographic composition of the general adult population in each country in which it is fielded, it is possible that the data may not be representative of the specific patient subpopulations examined in this study.

#### 9.10. Other Aspects

Not applicable.

#### 10. PROTECTION OF HUMAN PARTICIPANTS

#### 10.1. Patient Information

This study involves data that exist in deidentified/anonymized structured format and contain no patient personal information.

#### 10.2. Patient Consent

As this study involves deidentified/anonymized structured data, which according to applicable legal requirements do not contain data subject to privacy laws, obtaining informed consent from patients by Pfizer is not required.

#### 10.3. Institutional Review Board (IRB)/ Independent Ethics Committee (IEC)

IRB/IEC is not required for this study. However, the protocols and questionnaire associated with the original fielding of the 2023 US NHWS were reviewed by Pearl Institutional Review Board (Indianapolis, IN; Protocol Number: 2023-0121) and granted exemption from expedited or full ethical review. The granted exemption is stored on the Oracle server.

#### 10.4. Ethical Conduct of the Study

The study will be conducted in accordance with legal and regulatory requirements, as well as with scientific purpose, value, and rigor and follow generally accepted research practices described in Good Practices for Outcomes Research issued by the International Society for Pharmacoeconomics and Outcomes Research (ISPOR)<sup>18</sup>.

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

This study involves data that exist as structured data by the time of study start. In these data sources, individual patient data are not retrieved or validated, and it is not possible to link (i.e., identify a potential association between) a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event (AE) (i.e., identifiable patient, identifiable reporter, a suspect product, and event) cannot be met.

#### 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

Study results will be disseminated in the form of abstract submissions and poster presentations at the American Academy of Neurology (AAN) meeting in May 2025. For all publications relating to the study, Pfizer will comply with recognized ethical standards concerning publications and authorship.

In the event of any prohibition or restriction imposed (e.g., clinical hold) by an applicable competent authority in any area of the world, or if the party responsible for collecting data from the participant (i.e., Oracle Life Sciences) is aware of any new information which might influence the evaluation of the benefits and risks of a Pfizer product, Pfizer should be informed immediately.

#### 13. REFERENCES

- 1. Yang C, Liang C, Chang C, et al. Comparison of New Pharmacologic Agents With Triptans for Treatment of Migraine: A Systematic Review and Meta-analysis. JAMA Netw Open. 2021;4(10):e2128544. doi:10.1001/jamanetworkopen.2021.28544
- 2. Cameron C, Kelly S, Hsieh SC, Murphy M, Chen L, Kotb A, Peterson J, Coyle D, Skidmore B, Gomes T, Clifford T, Wells G. Triptans in the Acute Treatment of Migraine: A Systematic Review and Network Meta-Analysis. Headache. 2015 Jul-Aug;55 Suppl 4:221-35. doi: 10.1111/head.12601. Epub 2015 Jul 14. PMID: 26178694.
- 3. González-Hernández, A., Marichal-Cancino, B. A., MaassenVanDenBrink, A., & Villalón, C. M. (2018). Side effects associated with current and prospective antimigraine pharmacotherapies. Expert Opinion on Drug Metabolism & Toxicology, 14(1), 25–41. https://doi.org/10.1080/17425255.2018.1416097
- 4. Scott LJ. Rimegepant: First Approval. Drugs. 2020 May;80(7):741-746. doi: 10.1007/s40265-020-01301-3. PMID: 32270407.
- Blair HA. Rimegepant: A Review in the Acute Treatment and Preventive Treatment of Migraine. CNS Drugs. 2023 Mar;37(3):255-265. doi: 10.1007/s40263-023-00988-8.
   Epub 2023 Feb 4. Erratum in: CNS Drugs. 2023 Jul;37(7):661. PMID: 36739335; PMCID: PMC10299922.

- 6. DeFalco AP, Lazim R, Cope NE. Rimegepant Orally Disintegrating Tablet for Acute Migraine Treatment: A Review. Annals of Pharmacotherapy. 2021;55(5):650-657. doi:10.1177/1060028020954800
- 7. Lipton RB, Blumenfeld A, Jensen CM, Croop R, Thiry A, L'Italien G, Morris BA, Coric V, Goadsby PJ. Efficacy of rimegepant for the acute treatment of migraine based on triptan treatment experience: Pooled results from three phase 3 randomized clinical trials. Cephalalgia. 2023 Feb;43(2):3331024221141686. doi: 10.1177/03331024221141686. PMID: 36739511.
- 8. Buse DC, Rupnow MF, Lipton RB (2009) Assessing and managing all aspects of migraine: migraine attacks, migraine-related functional impairment, common comorbidities, and quality of life. Mayo Clin Proc 84:422–435
- 9. Bigal ME, Lipton RB (2009) The epidemiology, burden, and comorbidities of migraine. Neurol Clin 27:321–334
- Lombard, L., Farrar, M., Ye, W. et al. A global real-world assessment of the impact on health-related quality of life and work productivity of migraine in patients with insufficient versus good response to triptan medication. J Headache Pain 21, 41 (2020). https://doi.org/10.1186/s10194-020-01110-9
- 11. L'Italien G, Popoff E, Johnston K, et al. Rimegepant 75 mg for acute treatment of migraine is associated with significant reduction in monthly migraine days: Results from a long-term, open-label study. Cephalalgia Reports. 2022;5. doi:10.1177/25158163221075596
- 12. Johnston, K., Harris, L., Powell, L. et al. Monthly migraine days, tablet utilization, and quality of life associated with Rimegepant post hoc results from an open label safety study (BHV3000–201). J Headache Pain 23, 10 (2022). https://doi.org/10.1186/s10194-021-01378-5
- 13. Hays RD, Morales LS. The RAND-36 measure of health-related quality of life. Ann Med. 2001;33(5):350-357.
- 14. Herdman M, Gudex C, Lloyd A, et al. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qua Life Res. 2011;20(10):1727-1736.
- 15. Reilly MC, Arthur S. Zbrozek, Ellen M. Dukes. The validity and reproducibility of a work productivity and activity impairment instrument. Pharmacoeconomics. 1993;4(5):353-365.
- 16. Stewart, W. F., Lipton, R. B., Dowson, A. J., & Sawyer, J. (2001). Development and testing of the Migraine Disability Assessment (MIDAS) Questionnaire to assess headache-related disability. Neurology, 56(suppl 1), S20-S28.

- 17. Austin, P. C., & Stuart, E. A. (2015). Moving towards best practice when using inverse probability of treatment weighting (IPTW) using the propensity score to estimate causal treatment effects in observational studies. Statistics in medicine, 34(28), 3661-3679.
- 18. ISPOR. (2024). Good Practices Reports & More. Retrieved April 29, 2024, from https://www.ispor.org/heor-resources/good-practices.

#### 14. LIST OF TABLES

| Table 1. | Study Variables | .11 |
|----------|------------------------|-----|
| Table 2. | Estimated Sample Sizes | .14 |

#### 15. LIST OF FIGURES

Not applicable.

#### ANNEX 1. LIST OF STANDALONE DOCUMENTS

None.

#### **ANNEX 2. ADDITIONAL INFORMATION**

Not applicable.

## **Document Approval Record**

Document Name: C4951076\_NIS Protocol\_V1.0\_04Oct2024

**Document Title:** C4951076\_NIS Protocol\_V1.0\_04Oct2024

| Signed By: | Date(GMT) | Signing Capacity |
|------------|----------------------|------------------|
| PPD | 10-Oct-2024 13:59:50 | Manager Approval |